CLINICAL TRIAL: NCT00000877
Title: Steady-State Pharmacokinetic Interaction Study of Indinavir and Rifabutin
Brief Title: Study of How Indinavir (an Anti-HIV Drug) and Rifabutin (a Drug Used to Treat MAC, an HIV-Associated Disease) Interact in HIV-Positive and HIV-Negative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 365; 11328 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Rifabutin; Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; HIV Seronegativity; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Rifabutin

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Rifabutin

SUMMARY:
The purpose of this study is to evaluate the safety of giving indinavir and rifabutin at the same time (simultaneously) vs 4 hours apart (staggered) to HIV-positive and HIV-negative adults.

It is important to determine which medications for HIV-associated diseases, such as Mycobacterium avium complex (MAC) disease, can be given safely and effectively with anti-HIV drugs. Indinavir and rifabutin have been given simultaneously in the past with good results. This study seeks to examine if staggering the doses will make the 2 drugs more effective. HIV-negative volunteers are used in this study to examine the effect of rifabutin on indinavir and the effect of staggered rifabutin doses. The effect of rifabutin on the drug activity of indinavir is evaluated in HIV-positive patients.

DETAILED DESCRIPTION:
Currently, rifabutin is the only rifamycin that can be administered with indinavir. ACTG 365 is the first formal study of the pharmacokinetics of this dosing combination regimen in HIV seropositive patients. It is hypothesized that staggered administration of rifabutin and indinavir might minimize their pharmacokinetic interaction. If the intestinal tract plays a significant role in the presystemic clearance of rifabutin, the inhibitory activity of indinavir on rifabutin could depend on either luminal concentrations of indinavir, systematic concentrations of indinavir, or both. If luminal concentrations are important, then the interaction between these 2 drugs will be maximal when administered simultaneously, and minimal when their oral administration is staggered. Finally, since indinavir has a half-life of 1.8 hours, its effects on rifabutin's systematic clearance may be much less when administration of these drugs is staggered by 4 hours as compared with simultaneous administration with rifabutin. If the interaction on rifabutin is minimized, then the rifabutin levels may be suboptimal for treatment of tuberculosis in patients who are not administered the 2 drugs simultaneously. It is, therefore, important to define the magnitude of the effect of staggered vs simultaneous drug administration in order to clarify dose and regimen recommendations in HIV-infected patients with tuberculosis who also require protease inhibitor therapy.

Study Arm A is a multiple-dose, 3-period, sequential study in 18 evaluable HIV-infected indinavir-naive male and female volunteers [AS PER AMENDMENT 11/16/98: Arm A will be assessed in 18 evaluable HIV-seronegative patients]. Patients receive 3 different treatments consisting of 14 days of administration: rifabutin alone (Period IA); indinavir plus rifabutin (Period IIA); and indinavir plus rifabutin (Period IIIA). Study Arm B is a multiple-dose, 2-period, sequential study in 10 evaluable HIV-infected male and female volunteers. Patients receive 2 different treatments, each consisting of 14 days of administration; indinavir alone (Period IB); and indinavir plus rifabutin (Period IIB). Patients on both arms take each dose of their study medications with water. [AS PER AMENDMENT 8/8/97: Patients treated on Arm A are randomized, following Period IA therapy, to Period IIA or IIIA therapy for 14 days, then are crossed over to the alternate regimen for 14 days.] [AS PER AMENDMENT 4/17/98: After completion of therapy on Arm A or B, patients continue therapy with indinavir alone for 7 days.] [AS PER AMENDMENT 11/16/98: The final 7 days of indinavir dosing has been eliminated for patients on Arm A. Also per this amendment, to ensure compliance, Arm A patients' rifabutin supply will be dispensed in containers fitted with an electronic monitoring cap device.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive or HIV-negative.
* Agree to practice abstinence or to use birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have an active opportunistic (HIV-associated) disease or other disease requiring medication within 14 days of study entry.
* Have a history of illness that might put you at risk if given either of the study drugs.
* Have had any severe allergies to any substance in the past.
* Have a history of kidney stones.
* Have a medical condition, or problems with use of alcohol or drugs, which would keep you from completing the study.
* Have had tuberculosis and have never been treated for it.
* Are pregnant or breast-feeding.
* Are taking certain medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31
Dates: Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Flexner, Study Chair; Constance Benson, Study Chair; Judith Currier, Study Chair
Locations (8):
- United States (8):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of Southern California / LA County USC Med Cntr, Los Angeles, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York

REFERENCES:
- [Background] Hamzeh FM, Benson C, Gerber J, Currier J, McCrea J, Deutsch P, Ruan P, Wu H, Lee J, Flexner C; AIDS Clinical Trials Group 365 Study Team. Steady-state pharmacokinetic interaction of modified-dose indinavir and rifabutin. Clin Pharmacol Ther. 2003 Mar;73(3):159-69. doi: 10.1067/mcp.2003.3. PMID 12621381
- [Derived] Hennig S, Svensson EM, Niebecker R, Fourie PB, Weiner MH, Bonora S, Peloquin CA, Gallicano K, Flexner C, Pym A, Vis P, Olliaro PL, McIlleron H, Karlsson MO. Population pharmacokinetic drug-drug interaction pooled analysis of existing data for rifabutin and HIV PIs. J Antimicrob Chemother. 2016 May;71(5):1330-40. doi: 10.1093/jac/dkv470. Epub 2016 Jan 31. PMID 26832753